CLINICAL TRIAL: NCT05576246
Title: Airway Occlusion Measured During Non-invasive Ventilation to Assess Respiratory Effort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Olivos SMG (Other)
Collaborators: Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Principal Investigator, Marina Busico, Principal Investigator, Clinica Olivos SMG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Airway occlusion V1
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: non invasive ventilation; occlusion airway pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oclussion pressure (Experimental): The intervention consisted of measuring the esophageal pressure delta using an esophageal balloon (MBMed®). Once the balloon was placed and its correct position verified, NIV was initiated in three different scenarios (see procedure - NIV scenarios) in a randomized sequence, with allocation determined by sealed envelopes. During each scenario, ΔPocc was measured on the ventilator using an expiratory hold (3 measurements per scenario), and a stabilization period of 10 minutes was established before moving on to the next scenario.
  Interventions: Diagnostic Test: airway pressure occlusion measurement

INTERVENTIONS:
Diagnostic Test: airway pressure occlusion measurement — Flow, airway pressure (Paw), and esophageal pressure (Pes) will be recorded for 10 minutes on different NIV settings: during each one, three end-expiratory airway occlusions will be applied at random intervals. Each occlusion was maintained for the duration of a single breath deflection in Paw from PEEP, confirmed by the return of Paw to baseline.

SUMMARY:
Non-invasive ventilation (NIV) is extensively used in critical care settings and emergency departments for a variety of aetiologies but specially for acute respiratory failure (ARF). It eliminates morbidity related to the endotracheal tube and use of sedatives so it reduces intensive care unit (ICU) complications; however, on the other hand, the harmful effects of spontaneous breathing through the intensity of inspiratory effort may predispose the patient to the onset of self-inflicted lung injury (SILI). Therefore, measuring the level of inspiratory effort is recommended.The aim of this proof-of-concept physiological study was to describe the correlation between ΔPocc measured on the ventilator and ΔPes in healthy subjects with NIV.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is extensively used in critical care settings and emergency departments for a variety of aetiologies but specially for acute respiratory failure (ARF). Recommendations based on the GRADE methodology were addressed on several conditions such as exacerbation of chronic obstructive pulmonary disease (COPD), cardiogenic pulmonary oedema, de novo hypoxaemic respiratory failure, immunocompromised patients, chest trauma, palliative care, post-operative care, weaning and post-extubation period. NIV eliminates morbidity related to the endotracheal tube and use of sedatives so it reduces intensive care unit (ICU) acquired pneumonia, diaphragmatic atrophy, ICU acquired weakness and delirium. On the other hand, the harmful effects of spontaneous breathing through the intensity of inspiratory effort may follow a critical increase in respiratory drive, thus producing uncontrolled tidal change in dynamic transpulmonary pressure (PLdyn) that would increase the risk of injury to the dependent lung and predispose the patient to the onset of self-inflicted lung injury (SILI). High positive end-expiratory pressure (PEEP) renders spontaneous effort non injurious. P-SILI may worsen the clinical outcome of patients who require endotracheal intubation after having received noninvasive respiratory support. The underlying mechanisms of SILI are heterogeneous and include the pendelluft phenomenon, increased transvascular pressure gradient aggravating alveolar damage, excessive diaphragmatic loading with impaired systemic oxygen delivery and muscle injury. Therefore, measuring the level of inspiratory effort is recommended.

Esophageal manometry is a precise estimate of the changes in pleural pressure and is considered the gold standard to measure respiratory effort. Tonelli et al. measured tidal change in esophageal pressure (ΔPes) in patients with acute hypoxic de novo respiratory failure on NIV and demonstrated a median baseline value of ΔPes of 34 cmH2O that was significantly reduced within the first 2 hours of ventilation in patients who were successful in the NIV trial, whereas those failing the NIV trial did not show a significant reduction. However, esophageal manometry is rarely available bedside in acute settings on severe patients with respiratory distress so other ways of measuring inspiratory effort have been assessed, such as nasal pressure swings or the patient's respiratory effort against the occluded airway (ΔPocc). The latest was demonstrated on invasive mechanical ventilation patients. Lopez Navas et al. tried to correlate the inspiratory pressure-time product (PTPinsp) from transdiaphragmatic pressure to a novel expiratory occlusion method of 0.2 s in healthy volunteers with NIV on different settings; however, their results through Bland-Altman analysis of PTPinsp revealed mean differences between -4.22 and 7.57 cmH2O (SD 0.77- 8.52) and considerable differences between subjects. Moreover, Dargent A, et al. explored the feasibility of a noninvasive respiratory drive evaluation using ventilator-derived data as P0.1, clinical information and diaphragm ultrasound in COVID 19 patients on CPAP session with 5 cmH2O. They showed that P0.1 was achievable during NIV with a median value of 4.4 [2.7-5.1] cmH2O and not correlated with leaks, though they were small (5 [4-7] l/min); nevertheless, P0.1 was not accurate at predicting the risk of intubation but it was limited by its small sample size. In addition, P0.1 has been previously evaluated (with other physiological parameters) on NIV in COPD patients to predict post-extubation respiratory distress. They reported that only P0.1 recorded 1 h after the discontinuation of mechanical ventilation followed by 30 minutes of 4 cmH2O pressure support ventilation, was significantly different between the patients with and without respiratory distress (4.2 vs 1.8, p < 0.01). Nonetheless, there are no studies that measured bedside the pressure generated by the respiratory muscles during NIV.

The aim of this proof-of-concept physiological study was to describe the correlation between ΔPocc measured on the ventilator and ΔPes in healthy subjects with NIV.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects over 18 years old who wish to participate were included.

Exclusion Criteria:

* Exclusion criteria was the presence of any esophageal disease or COPD.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
correlation between ΔPocc measured on the ventilator and ΔPes in healthy subjects with NIV. | The subjects will be measured on each ventilator setting (3 settings) for 10 minutes
  Evaluate the agreement between ΔPocc and ΔPes in occluded breaths

SECONDARY OUTCOMES:
Correlation between Pccvent and PTPmus | The subjects will be measured on each ventilator setting (3 settings) for 10 minutes.
  The secondary outcome was the correlation between ΔPoccvent the mean PTPmus during the last minute of ventilation for each ventilator setting.
Correlation between Poccvent and Pesflux | The subjects will be measured on each ventilator setting (3 settings) for 10 minutes.
  Evaluate the agreement between ΔPocc and ΔPes in occluded breaths
  Evaluate the agreement between ΔPocc and ΔPes in non-occluded breaths
  Evaluate this relationship considering leak
  Evaluate the agreement between ΔPocc and PTPmin

CONTACTS AND LOCATIONS:
Overall Officials: Marina Busico, RT, Principal Investigator — Argentine Society of Intensive Care
Locations (1):
- Swiss Medical Group, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
we will intend to share our excel with the information af participant´s measurements so as to permit new hypothesis from other researchers

REFERENCES:
- [Result] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Result] Morais CCA, Koyama Y, Yoshida T, Plens GM, Gomes S, Lima CAS, Ramos OPS, Pereira SM, Kawaguchi N, Yamamoto H, Uchiyama A, Borges JB, Vidal Melo MF, Tucci MR, Amato MBP, Kavanagh BP, Costa ELV, Fujino Y. High Positive End-Expiratory Pressure Renders Spontaneous Effort Noninjurious. Am J Respir Crit Care Med. 2018 May 15;197(10):1285-1296. doi: 10.1164/rccm.201706-1244OC. PMID 29323536
- [Result] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. Spontaneous breathing during lung-protective ventilation in an experimental acute lung injury model: high transpulmonary pressure associated with strong spontaneous breathing effort may worsen lung injury. Crit Care Med. 2012 May;40(5):1578-85. doi: 10.1097/CCM.0b013e3182451c40. PMID 22430241
- [Result] Grieco DL, Menga LS, Eleuteri D, Antonelli M. Patient self-inflicted lung injury: implications for acute hypoxemic respiratory failure and ARDS patients on non-invasive support. Minerva Anestesiol. 2019 Sep;85(9):1014-1023. doi: 10.23736/S0375-9393.19.13418-9. Epub 2019 Mar 12. PMID 30871304
- [Result] Battaglini D, Robba C, Ball L, Silva PL, Cruz FF, Pelosi P, Rocco PRM. Noninvasive respiratory support and patient self-inflicted lung injury in COVID-19: a narrative review. Br J Anaesth. 2021 Sep;127(3):353-364. doi: 10.1016/j.bja.2021.05.024. Epub 2021 Jun 3. PMID 34217468
- [Result] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. The comparison of spontaneous breathing and muscle paralysis in two different severities of experimental lung injury. Crit Care Med. 2013 Feb;41(2):536-45. doi: 10.1097/CCM.0b013e3182711972. PMID 23263584
- [Result] Gainnier M, Roch A, Forel JM, Thirion X, Arnal JM, Donati S, Papazian L. Effect of neuromuscular blocking agents on gas exchange in patients presenting with acute respiratory distress syndrome. Crit Care Med. 2004 Jan;32(1):113-9. doi: 10.1097/01.CCM.0000104114.72614.BC. PMID 14707568
- [Result] Telias I, Spadaro S. Techniques to monitor respiratory drive and inspiratory effort. Curr Opin Crit Care. 2020 Feb;26(1):3-10. doi: 10.1097/MCC.0000000000000680. PMID 31764192
- [Result] Tonelli R, Fantini R, Tabbi L, Castaniere I, Pisani L, Pellegrino MR, Della Casa G, D'Amico R, Girardis M, Nava S, Clini EM, Marchioni A. Early Inspiratory Effort Assessment by Esophageal Manometry Predicts Noninvasive Ventilation Outcome in De Novo Respiratory Failure. A Pilot Study. Am J Respir Crit Care Med. 2020 Aug 15;202(4):558-567. doi: 10.1164/rccm.201912-2512OC. PMID 32325004
- [Result] Tonelli R, Cortegiani A, Marchioni A, Fantini R, Tabbi L, Castaniere I, Biagioni E, Busani S, Nani C, Cerbone C, Vermi M, Gozzi F, Bruzzi G, Manicardi L, Pellegrino MR, Beghe B, Girardis M, Pelosi P, Gregoretti C, Ball L, Clini E. Nasal pressure swings as the measure of inspiratory effort in spontaneously breathing patients with de novo acute respiratory failure. Crit Care. 2022 Mar 24;26(1):70. doi: 10.1186/s13054-022-03938-w. PMID 35331323
- [Result] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692
- [Result] Lopez-Navas K, Brandt S, Strutz M, Gehring H, Wenkebach U. Non-invasive determination of respiratory effort in spontaneous breathing and support ventilation: a validation study with healthy volunteers. Biomed Tech (Berl). 2014 Aug;59(4):335-41. doi: 10.1515/bmt-2013-0057. PMID 24607917
- [Result] Dargent A, Hombreux A, Roccia H, Argaud L, Cour M, Guerin C. Feasibility of non-invasive respiratory drive and breathing pattern evaluation using CPAP in COVID-19 patients. J Crit Care. 2022 Jun;69:154020. doi: 10.1016/j.jcrc.2022.154020. Epub 2022 Mar 17. PMID 35306443
- [Result] Hilbert G, Gruson D, Portel L, Vargas F, Gbikpi-Benissan G, Cardinaud JP. Airway occlusion pressure at 0.1 s (P0.1) after extubation: an early indicator of postextubation hypercapnic respiratory insufficiency. Intensive Care Med. 1998 Dec;24(12):1277-82. doi: 10.1007/s001340050762. PMID 9885880
- [Result] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443